CLINICAL TRIAL: NCT01323660
Title: An Exercise Endurance Study to Evaluate the Effects of Treatment of Chronic Obstructive Pulmonary Disease (COPD) Patients With a Dual Bronchodilator: GSK573719/GW642444. Study B
Brief Title: An Exercise Endurance Study to Evaluate the Effects of Treatment of Chronic Obstructive Pulmonary Disease (COPD) Patients With a Dual Bronchodilator: GSK573719/GW642444.Study B
Acronym: COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 114418
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- GSK573719/GW642444 125/25 (Experimental): 125mcg/25mcg nDPI
  Interventions: Drug: GSK573719 125; Drug: GW642444 25; Device: placebo
- GSK573719/GW642444 62.5/25 (Experimental): 62.5mcg/25mcg nDPI
  Interventions: Drug: GSK573719 62.5; Drug: GW642444 25; Device: placebo
- GSK573719/ 125 (Experimental): 125mcg nDPI
  Interventions: Drug: GSK573719/GW642444 125/25; Device: placebo
- GSK573719 62.5 (Experimental): 62.5mcg nDPI
  Interventions: Drug: GSK573719/GW642444 62.5/25; Device: placebo
- GW642444 25 (Experimental): 25mcg nDPI
  Interventions: Drug: GSK573719/GW642444 125/25; Drug: GSK573719/GW642444 62.5/25; Device: placebo
- Placebo (Placebo Comparator): Plb nDPI
  Interventions: Drug: GSK573719/GW642444 125/25; Drug: GSK573719/GW642444 62.5/25; Drug: GSK573719 125; Drug: GSK573719 62.5; Drug: GW642444 25

INTERVENTIONS:
Drug: GSK573719/GW642444 125/25 — 125mcg/ 25mcg QID (Once daily , inhaled)
  Arms: GSK573719/ 125; GW642444 25; Placebo
Drug: GSK573719/GW642444 62.5/25 — 62.5mcg/25mcg QID
  Arms: GSK573719 62.5; GW642444 25; Placebo
Drug: GSK573719 125 — 125mcg QID
  Arms: GSK573719/GW642444 125/25; Placebo
Drug: GSK573719 62.5 — 62.5mcg QID
  Arms: GSK573719/GW642444 62.5/25; Placebo
Drug: GW642444 25 — 25mcg QID
  Arms: GSK573719/GW642444 125/25; GSK573719/GW642444 62.5/25; Placebo
Device: placebo — Comparator QID
  Arms: GSK573719 62.5; GSK573719/ 125; GSK573719/GW642444 125/25; GSK573719/GW642444 62.5/25; GW642444 25

SUMMARY:
This is a phase III multicenter, randomized, double-blind, placebo-controlled, combination and component, two-period, incomplete block design cross-over study using GSK573719/GW642444. The primary objective is to evaluate lung function and exercise endurance time after 12 weeks of once-daily administration of GSK573719/GW642444 Inhalation Powder (125/25mcg and 62.5/25mcg), GSK573719 Inhalation Powder (125mcg and 62.5mcg), GW642444 Inhalation Powder 25 mcg and placebo delivered by a Novel dry powder inhaler (Novel DPI).

DETAILED DESCRIPTION:
Expiratory airflow limitation is the most obvious physiological change associated with chronic obstructive pulmonary disease (COPD). A consequence of airflow limitation is gas trapping as expiration becomes flow limited. This may occur at rest with more severe airway obstruction and is most evident during exercise as lung emptying is reduced and increased ventilation does not allow full expiration. This increased gas trapping or hyperinflation is the cause of much of the increased work of breathing, dyspnea, and exercise intolerance in subjects with COPD (O'Donnell 1997; O'Donnell, 1993). Spirometric measurement of airflow limitation, particularly as assessed by forced expiratory volume in one second (FEV1), is commonly used for the diagnosis of and assessment of response to pharmacotherapeutic intervention in COPD. However, changes in FEV1 may not fully predict symptomatic responses and alternative measures of lung hyperinflation such as exercise tolerance and exertional dyspnea may be more sensitive to therapeutic intervention and/or more clinically relevant than FEV1 [O'Donnell1999; Bauerle, 1998; O'Donnell, 1998; Officer, 1998]. GSK573719/GW642444 Inhalation Powder, a combination of the long-acting muscarinic antagonist (LAMA) bronchodilator GSK573719 and the long-acting beta2-agonist (LABA) bronchodilator GW642444, is in development for the maintenance treatment of airflow obstruction associated with COPD. Development of this product is supported by studies showing improvement in lung function with similar safety when use of combinations of long-acting bronchodilators with different mechanisms of action are compared with single bronchodilator therapy [van Noord 2005; van Noord van Noord 2006; Tashkin 2008]. Previous studies have demonstrated that treatment with short- and long-acting bronchodilators including ipratropium, tiotropium, and salmeterol reduces resting lung hyperinflation as measured by functional residual capacity (FRC), residual volume (RV), and inspiratory capacity (IC), with associated improvements in exercise endurance time and exertional dyspnoea in subjects with COPD [Ayers, 2001; O'Donnell 1998; O'Donnell 2004; Pepin 2005; Pepin 2007; Ramirez-Venegas 1997]. However, the effect of combined LAMA/LABA therapy on these measures is not well characterized.

This is a phase III multicenter, randomized, double-blind, placebo-controlled, combination and component, two-period, incomplete block design cross-over study using GSK573719/GW642444. The primary objective is to evaluate lung function and exercise endurance time after 12 weeks of once-daily administration of GSK573719/GW642444 Inhalation Powder (125/25mcg and 62.5/25mcg), GSK573719 Inhalation Powder (125mcg and 62.5mcg), GW642444 Inhalation Powder 25 mcg and placebo delivered by a Novel dry powder inhaler (Novel DPI) Approximately 312 subjects with moderate/severe chronic obstructive pulmonary disease (COPD) will be randomised in order to achieve 208 subjects completing both treatment periods of 3 months.. There will be a total of 12 study clinic visits conducted on an outpatient basis. Subjects who meet the eligibility criteria at Screening (Visit 1) will complete a 12 to 21 day run-in period followed by two 12-week treatment periods that are separated by a 14 day wash-out. Clinic visits will be conducted at Screening (Visit 1), twice during the run-in period (Visits 2 and 3), at randomization (Visit 4) and three times during the first treatment period, on Treatment Day 2 (Visit 5) and at 6 and 12 weeks (Visits 6 and 7 respectively). During the washout period of 14 days there will be 2 clinic visits (Visits 8 and 9). During the second treatment period there will be 3 clinic visits, on Treatment Day 2 (Visit 10) and at 6 and 12 weeks (Visits 11 and 12 respectively). A Safety Follow-Up assessment (Visit 13) to record adverse events will be conducted by telephone 7 days after the end of the second treatment period or early withdrawal. Efficacy measurements will include pre and post dose FEV1, lung volume measurements and exercise endurance time measured using the endurance shuttle walking test (ESWT). Safety and tolerability will be assessed by collection of adverse events (AEs), vital signs, 12-lead electrocardiograms (ECGs), clinical laboratory tests and incidence of COPD exacerbations. Dyspnea will be assessed using the Exercise Dyspnea Scale (EDS), a patient-reported outcome. Blood samples will also be collected for potential pharmacogenetics analysis

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: 40 years of age or older at Visit 1.
* Gender: Male or female subjects.
* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society [Celli, 2004]
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of ≥ 10 pack-years
* Severity of Disease: A post-albuterol/salbutamol FEV1/FVC ratio of 0.70 and a post-albuterol/salbutamol FEV1 of >35% and <70% of predicted normal
* Dyspnea: A score of ≥2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Visit 1
* Resting Lung Volumes: A resting FRC of ≥120% of predicted normal FRC at Visit 1.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known respiratory disorders other than COPD including but not limited to alpha-1 antitrypsin deficiency, active tuberculosis, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, and interstitial lung disease. Allergic rhinitis is not exclusionary.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for < 5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study. Any physical or mental abnormality which would affect the patient carrying out exercise tests including peripheral vascular disease should be excluded at the investigators discretion.
* Chest X-Ray: A chest X-ray or computed tomography (CT) scan that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken at Visit 1 if a chest X-ray or CT scan is not available within 6 months prior to Visit 1. For subjects in Germany, if a chest X-ray (or CT scan) is not available in the 6 months prior to Visit 1 the subject will not be eligible for the study.
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* 12-Lead ECG: An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1, including the presence of a paced rhythm on a 12-lead electrocardiogram (ECG) which causes the underlying rhythm and ECG to be obscured. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility.
* Screening Labs: Significantly abnormal finding from clinical chemistry and hematology tests at Visit 1.
* Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications prior to Screening, including depot,oral corticosteroids, combinations of LABA/ICS, LABA, PDE4 inhibitors.
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulized therapy
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2011-03-16; Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (18):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Livonia, Michigan
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Richmond, Virginia
- Canada (4):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Czechia (5):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Karlovy Vary
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Teplice
- Denmark (4):
  - GSK Investigational Site, Aarhus C
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, København NV
  - GSK Investigational Site, Odense C
- South Africa (6):
  - GSK Investigational Site, George, Eastern Cape
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Groenkloof
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Panorama
- Ukraine (3):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
- United Kingdom (9):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Cottingham, East Yorkshire
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Somerset
  - GSK Investigational Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) who were eligible completed a 12- to 21-day Run-in Period followed by two 12-week treatment (trt) periods.
Pre-assignment Details: A total of 634 par. were enrolled and screened, 393 par. entered the Run-in Period, 308 par. were randomized and 307 par. received study trt. Participant Flow data are presented by treatment rather than sequence. Par. received 2 out of the 6 interventions.
Groups:
- Placebo: Participants received matching placebo once daily (QD) via a dry powder inhaler (DPI) in the morning for 12weeks.
- UMEC 62.5 µg QD: Participants received umeclidinium bromide (UMEC) 62.5 micrograms (µg) QD via a DPI in the morning for 12 weeks.
- UMEC 125 µg QD: Participants received UMEC 125 µg QD via a DPI in the morning for 12 weeks.
- VI 25 µg QD: Participants received vilanterol (VI) 25 µg QD via a DPI for 12 weeks.
- UMEC/VI 62.5/25 µg QD: Participants received UMEC/VI 62.5/25 µg QD via a DPI in the morning for 12 weeks.
- UMEC 125/25 µg QD: Participants received UMEC/VI 125/25 µg QD via a DPI in the morning for 12 weeks.
Period: Treatment Period 1 (12 Weeks)
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC 125/25 µg QD
Started | 84 | 22 | 24 | 36 | 71 | 70
Completed | 65 | 21 | 19 | 31 | 61 | 61
Not Completed | 19 | 1 | 5 | 5 | 10 | 9
Not completed — Adverse Event | 6 | 1 | 1 | 3 | 3 | 4
Not completed — Lack of Efficacy | 6 | 0 | 2 | 0 | 1 | 3
Not completed — Protocol Violation | 2 | 0 | 1 | 1 | 1 | 2
Not completed — Met Protocol-defined Stopping Criteria | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 1 | 1 | 3 | 0
Period: Washout Period (14 Days)
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC 125/25 µg QD
Started | 65 | 21 | 19 | 31 | 61 | 61
Completed | 65 (Participants withdrawing during washout are counted under the last treatment taken.) | 21 (Participants withdrawing during washout are counted under the last treatment taken.) | 18 (Participants withdrawing during washout are counted under the last treatment taken.) | 28 (Participants withdrawing during washout are counted under the last treatment taken.) | 58 (Participants withdrawing during washout are counted under the last treatment taken.) | 59 (Participants withdrawing during washout are counted under the last treatment taken.)
Not Completed | 0 | 0 | 1 | 3 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 3 | 2 | 2
Period: Treatment Period 2 (12 Weeks)
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC 125/25 µg QD
Started | 67 ("By crossover design, participants were assigned to a different treatment arm in each period.) | 18 ("By crossover design, participants were assigned to a different treatment arm in each period.) | 17 ("By crossover design, participants were assigned to a different treatment arm in each period.) | 28 ("By crossover design, participants were assigned to a different treatment arm in each period.) | 59 ("By crossover design, participants were assigned to a different treatment arm in each period.) | 58 ("By crossover design, participants were assigned to a different treatment arm in each period.)
Completed | 55 | 17 | 14 | 25 | 55 | 51
Not Completed | 12 | 1 | 3 | 3 | 4 | 7
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 1 | 2
Not completed — Lack of Efficacy | 9 | 0 | 2 | 2 | 1 | 3
Not completed — Study Closed/Terminated | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Treatments: Participants were randomized to receive a sequence consisting of 2 of the following treatments: UMEC/VI 125/25 µg , UMEC/VI 62.5/25 µg , UMEC 125 µg , UMEC 62.5 µg , VI 25 µg , or placebo QD via a DPI. Each treatment was administered in the morning for 12 weeks. The treatment periods were seperated by 14-day washout period.
Arm/Group | All Study Treatments
Number analyzed (Participants) | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 168
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 6
  American Indian or Alaska Native | 1
  Asian - South East Asian Heritage | 1
  White - White/Caucasian/European Heritage | 298
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Exercise Endurance Time Post-dose at Week 12 of Each Treatment Period
Description: Exercise endurance time (EET) post-dose at Week 12 is defined as the EET obtained 3 hours after dosing at Week 12. EET was measured using the externally paced field walking test called the endurance shuttle walk test (ESWT). Analysis performed using a repeated measures model with covariates of period walking speed, mean walking speed, period, treatment, visit, smoking status, center group, visit by period walking speed, visit by mean walking speed and visit by treatment interactions. The model used all available 3-hour post-dose change from baseline EET values recorded on Day 2, Week 6 and Week 12. Baseline was the EET assessment obtained prior to dosing on Day 1 of each period. The mean walking speed for each participant is the mean of the levels used for the ESWT in each of the two treatment periods. The period walking speed for each participant and treatment period is the difference between the level for that participant and period and the mean walking speed for that participant.
Time Frame: Week 12 of each treatment period (up to Study Week 30)
Population: Intent-to-Treat (ITT) Population: all par. randomized to treatment who received at least one dose of study drug in either treatment period. Number of par. represent those with data available at the time point; however, all par. in the ITT population without missing covariate information and with at least one post Baseline measurement are included.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Groups:
- Placebo: Participants received matching placebo QD via a DPI in the morning for 12 weeks.
- UMEC 62.5 µg QD: Participants received UMEC 62.5 µg QD via a DPI in the morning for 12 weeks.
- VI 25 µg QD: Participants received VI 25 µg QD via a DPI for 12 weeks.
- UMEC/VI 125/25 µg QD: Participants received UMEC/VI 125/25 µg QD via a DPI in the morning for 12 weeks.
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 117 | 37 | 32 | 54 | 115 | 109
Seconds | 0.1 (16.66) | 25.1 (30.18) | 74.8 (31.58) | 30.7 (24.79) | 69.5 (17.09) | 65.9 (17.48)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p = 0.456, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 25.0, 95% CI 2-sided [-41.0 to 91.0] — Least square mean change difference=UMEC 62.5 µg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs UMEC 125 µg QD; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 74.7, 95% CI 2-sided [6.0 to 143.4] — Least square mean change difference=UMEC 125 µg minus Placebo
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg QD; Test type: Superiority or Other; p = 0.295, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 30.6, 95% CI 2-sided [-26.8 to 88.0] — Least square mean change difference=VI 25 µg minus Placebo
Statistical Analysis 4: Comparison: UMEC 62.5 µg QD vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p = 0.188, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 44.4, 95% CI 2-sided [-21.8 to 110.6] — Least square mean change difference=UMEC/VI 62.5/25 µg minus UMEC 62.5 µg
Statistical Analysis 5: Comparison: VI 25 µg QD vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p = 0.187, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 38.8, 95% CI 2-sided [-18.9 to 96.5] — Least square mean change difference=UMEC/VI 62.5/25 µg minus VI 25 µg
Statistical Analysis 6: Comparison: UMEC 125 µg QD vs UMEC/VI 125/25 µg QD; Test type: Superiority or Other; p = 0.801, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = -8.9, 95% CI 2-sided [-77.8 to 60.1] — Least square mean change difference=UMEC/VI 125/25 µg minus UMEC 125 µg
Statistical Analysis 7: Comparison: VI 25 µg QD vs UMEC/VI 125/25 µg QD; Test type: Superiority or Other; p = 0.233, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 35.2, 95% CI 2-sided [-22.7 to 93.1] — Least square mean change difference=UMEC/VI 125/25 µg minus VI 25 µg
Statistical Analysis 8: Comparison: Placebo vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 69.4, 95% CI 2-sided [24.5 to 114.4] — Least square mean change difference=UMEC/VI 62.5/25 µg minus Placebo
Statistical Analysis 9: Comparison: Placebo vs UMEC/VI 125/25 µg QD; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 65.8, 95% CI 2-sided [20.3 to 111.3] — Least square mean change difference=UMEC/VI 125/25 µg minus Placebo

2. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Week 12 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry on Day 2, Week 6 and Week 12. Baseline is the FEV1 value recorded pre-dose on Day 1 of each treatment period, mean Baseline is the mean of the Baselines for each participant, and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Clinic visit trough (pre-bronchodilator and pre-dose) FEV1 at Week 12 (Treatment Day 85) is defined as the FEV1 value obtained 24 hours after dosing on Treatment Day 84. Analysis performed using a repeated measures model with covariates of period Baseline, mean Baseline, period, treatment, visit, smoking status, center group, visit by period Baseline, visit by mean Baseline and visit by treatment interactions.
Time Frame: Week 12 of each treatment period (up to Study Week 30)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 119 | 38 | 33 | 56 | 117 | 112
Liters | -0.043 (0.0156) | 0.101 (0.0267) | 0.212 (0.0287) | 0.069 (0.0222) | 0.200 (0.0156) | 0.218 (0.0159)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.144, 95% CI 2-sided [0.086 to 0.203] — Least square mean change difference=UMEC 62.5 µg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs UMEC 125 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.255, 95% CI 2-sided [0.193 to 0.318] — Least square mean change difference=UMEC 125 µg minus Placebo
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.112, 95% CI [0.061 to 0.163] — Least square mean change difference=VI 25 µg minus Placebo
Statistical Analysis 4: Comparison: UMEC 62.5 µg QD vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.099, 95% CI 2-sided [0.041 to 0.157] — Least square mean change difference=UMEC/VI 62.5/25 µg minus UMEC 62.5 µg
Statistical Analysis 5: Comparison: VI 25 µg QD vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.132, 95% CI 2-sided [0.081 to 0.183] — Least square mean change difference=UMEC/VI 62.5/25 µg minus VI 25 µg
Statistical Analysis 6: Comparison: UMEC 125 µg QD vs UMEC/VI 125/25 µg QD; Test type: Superiority or Other; p = 0.849, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.006, 95% CI 2-sided [-0.055 to 0.067] — Least square mean change difference=UMEC/VI 125/25 µg minus UMEC 125 µg
Statistical Analysis 7: Comparison: VI 25 µg QD vs UMEC/VI 125/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.150, 95% CI 2-sided [0.098 to 0.201] — Least square mean change difference=UMEC/VI 125/25 µg minus VI 25 µg
Statistical Analysis 8: Comparison: Placebo vs UMEC/VI 62.5/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.243, 95% CI 2-sided [0.202 to 0.284] — Least square mean change difference=UMEC/VI 62.5/25 µg minus Placebo
Statistical Analysis 9: Comparison: Placebo vs UMEC/VI 125/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.261, 95% CI 2-sided [0.220 to 0.303] — Least square mean change difference=UMEC/VI 125/25 µg minus Placebo

3. Secondary Outcome: Change From Baseline in Inspiratory Capacity (Trough and 3-hours Post-dose) at Week 12 of Each Treatment Period
Description: Inspiratory capacity (IC) is defined as the maximum amount of air that can be inhaled into the lungs from the normal resting position after breathing out normally. Baseline is the IC value recorded pre-dose on Day 1 of each treatment period, mean Baseline is the mean of the Baselines for each participant, and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Trough IC is measured pre-dose on Treatment Week 12 of each treatment period. IC 3-hours post-dose is measured from the value obtained 3 hours after dosing on Treatment Week 12 of each treatment period. Analysis performed using a repeated measures model with covariates of period Baseline, mean Baseline, period, treatment, visit, smoking status, center group, visit by period Baseline, visit by mean Baseline and visit by treatment interactions. IC measurements were taken electronically by plethysmography on Day 2, Week 6 and Week 12.
Time Frame: Week 12 of each treatment period (up to Study Week 30)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 120 | 38 | 33 | 56 | 117 | 111
Liters
  Trough | -0.021 (0.0271) | 0.077 (0.0471) | 0.216 (0.0505) | 0.081 (0.0391) | 0.216 (0.0274) | 0.204 (0.0281)
  3-hours post-dose | -0.021 (0.0273) | 0.155 (0.0465) | 0.208 (0.0498) | 0.156 (0.0389) | 0.295 (0.0276) | 0.312 (0.0283)

4. Secondary Outcome: Change From Baseline in Functional Residual Capacity (Trough and 3-hours Post-dose) at Week 12 of Each Treatment Period
Description: Functional Residual Capacity (FRC) is defined as the amount of air still left in the lungs after breathing out normally. Baseline is the FRC value recorded pre-dose on Day 1 of each treatment period, mean Baseline is the mean of the Baselines for each participant, and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Trough FRC is measured pre-dose on Treatment Week 12. FRC 3-hours post-dose is measured from the value obtained 3 hours after dosing on Treatment Week 12. Analysis performed using a repeated measures model with covariates of period Baseline, mean Baseline, period, treatment, visit, smoking status, center group, visit by period Baseline, visit by mean Baseline and visit by treatment interactions. FRC measurements were taken electronically by plethysmography on Day 2, Week 6 and Week 12.
Time Frame: Week 12 of each treatment period (up to Study Week 30)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 120 | 38 | 33 | 56 | 117 | 111
Liters
  Trough | -0.083 (0.0460) | -0.200 (0.0804) | -0.263 (0.0862) | -0.218 (0.0666) | -0.434 (0.0469) | -0.333 (0.0480)
  3-hours post-dose | -0.094 (0.0461) | -0.315 (0.0786) | -0.405 (0.0836) | -0.431 (0.0654) | -0.616 (0.0471) | -0.503 (0.0480)

5. Secondary Outcome: Change From Baseline in Residual Volume (Trough and 3-hours Post-dose) at Week 12 of Each Treatment Period
Description: Residual Volume (RV) is defined as the air that remains in the lungs after breathing out as fully as possible. Baseline is the RV value recorded pre-dose on Day 1 of each treatment period, mean Baseline is the mean of the Baselines for each participant, and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Trough RV is measured pre-dose on Treatment Week 12. RV 3-hours post-dose is measured from the value obtained 3 hours after dosing on Treatment Week 12. Analysis performed using a repeated measures model with covariates of period Baseline, mean Baseline, period, treatment, visit, smoking status, center group, visit by period Baseline, visit by mean Baseline and visit by treatment interactions. RV measurements were taken electronically by plethysmography on Day 2, Week 6 and Week 1.
Time Frame: Week 12 of each treatment period (up to Study Week 30)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 120 | 38 | 33 | 56 | 117 | 111
Liters
  Trough | -0.049 (0.0491) | -0.266 (0.0847) | -0.289 (0.0909) | -0.291 (0.0705) | -0.516 (0.0500) | -0.421 (0.0511)
  3-hours post-dose | -0.071 (0.0495) | -0.451 (0.0855) | -0.534 (0.0911) | -0.483 (0.0711) | -0.714 (0.0505) | -0.566 (0.0516)

6. Secondary Outcome: Change From Baseline in 3-hours Post-dose FEV1 at Week 12 of Each Treatment Period
Description: FEVI is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Baseline is the FEV1 value recorded pre-dose on Day 1 of each treatment period, mean Baseline is the mean of the Baselines for each participant, and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Clinic visit post-dose FEV1 at Week 12 (Treatment Day 85) is defined as the FEV1 value obtained 3 hours after dosing on Treatment Day 85. Analysis performed using a repeated measures model with covariates of period Baseline, mean Baseline, period, treatment, visit, smoking status, center group, visit by period Baseline, visit by mean Baseline and visit by treatment interactions 3 hour post-dose FEV1 measurements were taken electronically by spirometry on Day 2, Week 6 and Week 12.
Time Frame: Week 12 of each treatment period (up to Study Week 30)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Number analyzed (Participants) | 120 | 38 | 33 | 56 | 117 | 110
Liters | -0.019 (0.0175) | 0.168 (0.0296) | 0.215 (0.0317) | 0.143 (0.0246) | 0.297 (0.0175) | 0.343 (0.0179)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs), defined as those events occuring while participants were on treatment up until one day after the last dose (up to Week 33), are reported.
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | VI 25 µg QD | UMEC/VI 62.5/25 µg QD | UMEC/VI 125/25 µg QD
Serious Adverse Events (participants affected / at risk) | 4/151 | 1/40 | 1/41 | 2/64 | 3/130 | 5/128
Other Adverse Events (participants affected / at risk) | 31/151 | 5/40 | 14/41 | 12/64 | 20/130 | 18/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | UMEC 62.5 µg QD (N=40) | UMEC 125 µg QD (N=41) | VI 25 µg QD (N=64) | UMEC/VI 62.5/25 µg QD (N=130) | UMEC/VI 125/25 µg QD (N=128)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
IIIrd nerve paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | UMEC 62.5 µg QD (N=40) | UMEC 125 µg QD (N=41) | VI 25 µg QD (N=64) | UMEC/VI 62.5/25 µg QD (N=130) | UMEC/VI 125/25 µg QD (N=128)
Nasopharyngitis (Infections and infestations) | 10 | 4 | 4 | 1 | 8 | 2
Sinusitis (Infections and infestations) | 3 | 0 | 2 | 3 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Headache (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 4 | 1 | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 2 | 2 | 5
Dyspnoea (Gastrointestinal disorders) | 6 | 0 | 1 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.